CLINICAL TRIAL: NCT02038790
Title: A Single Center, Randomized, 2 Way Cross-Over, Phase 4 Study Comparing Usability of Zubsolv Sublingual Tablets 5.7/1.4 to Suboxone Sublingual Film 8/2 Including Ease of Use, Taste Preference, Dissolution Time, Desire to Abuse, and Overall Acceptance In Buprenorphine/Naloxone Treated Opioid Dependent Population
Brief Title: Usability of Zubsolv Sublingual Tablets 5.7/1.4 to Suboxone Sublingual Film 8/2 In Buprenorphine/Naloxone Treated Opioid Dependent Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RBP-OSZ1; 13-131220-108 (Other: Hill Top Research)
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; buprenorphine/naloxone; Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suboxone sublingual film 8/2 (Experimental): Participants took a single dose of Suboxone sublingual film 8/2 either on Day 0 or Day 1, depending on the how each participant was randomized in this cross-over study.
  Interventions: Drug: Suboxone Sublingual Film
- Zubsolv sublingual tablets 5.7/1.4 (Active Comparator): Participants took a single dose of Zubsolv sublingual tablets 5.7/1.4 either on Day 0 or Day 1, depending on the how each participant was randomized in this cross-over study.
  Interventions: Drug: Zubsolv sublingual tablets

INTERVENTIONS:
Drug: Suboxone Sublingual Film — A single Suboxone sublingual film strip containing 8mg buprenorphine and 2mg naloxone taken sublingually on either Day 0 or Day 1, depending on randomized treatment arm assignment. Study drug will be administered by designated qualified study personnel at the site in the morning prior to 9:00 a.m. under fasting conditions.
  Other Names: buprenorphine; naloxone
  Arms: Suboxone sublingual film 8/2
Drug: Zubsolv sublingual tablets — A single Zubsolv sublingual tablet containing 5.7mg buprenorphine and 1.4mg naloxone taken sublingually on either Day 0 or Day 1, depending on randomized treatment arm assignment. Study drug will be administered by designated qualified study personnel at the site in the morning prior to 9:00 a.m. under fasting conditions.
  Other Names: buprenorphine; naloxone
  Arms: Zubsolv sublingual tablets 5.7/1.4

SUMMARY:
The primary objective of this study is to compare overall patient preference for either Suboxone® sublingual film 8/2 or Zubsolv® sublingual tablets 5.7/1.4. Suboxone sublingual film 8/2 contains 8mg buprenorphine and 2mg naloxone. Zubsolv sublingual tablets contain 5.7 mg buprenorphine and 1.4 mg naloxone. Both interventions act as a substitute for opiate drugs like heroin, morphine or oxycodone and help withdrawal from opiate drugs over a period of time.

ELIGIBILITY:
Inclusion Criteria:

* currently on a single daily dose of 8/2 of Suboxone or generic equivalent, or 5.7/1.4 mg Zubsolv for treatment of opioid dependence that has been medically confirmed.
* in good general health with no specific contraindication for treatment with buprenorphine or naloxone.
* the ability to understand, sign and date written consent and Health Information Portability and Accountability Act (HIPAA) authorization forms, which must be obtained prior to any study related procedures being completed.
* Female subjects must be postmenopausal for at least 2 years, surgically sterile (i.e. tubal ligation, hysterectomy, or bilateral ovariectomy), or practicing an effective method of contraception during the study with one of the following methods: oral contraception, intrauterine device (IUD), abstinence, contraceptive injections, conscientious use of a diaphragm or condoms and spermicidal foam, systemic (implant) contraception or partner has had a vasectomy.

Exclusion Criteria:

* Subject is taking other opioids (other than buprenorphine/naloxone) that may interfere with the study evaluations or compromise the safety of the subject.
* Subject is not able to read or have other impairments that may prevent completion of questionnaires or other study evaluations
* Subject has open sores present in the oral cavity.
* Subject has participated in any previous clinical testing involving investigational drug within the 4 weeks prior to study start.
* Subject is pregnant, lactating or planning a pregnancy
* Subject is currently participating in any other type of clinical testing.
* Subject has a medical condition that in the Investigator's opinion could affect the taste assessments required by the study
* Subject is judged by the Investigator after reviewing medical history to be unsuitable for any other reason that may either place the subject at increased risk during participation or interfere with the interpretation of the study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Murray, MD, Principal Investigator — Hill Top Research
Locations (1):
- Hill Top Research, St. Petersburg, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty nine (39) subjects were screened and thirty three (33) subjects were enrolled in the study.
Groups:
- Suboxone - Zubsolv: Participants received Suboxone® (buprenorphine 8 mg /naloxone 2 mg sublingual film) on Day 0 and Zubsolv® (buprenorphine 5.7 mg /naloxone 1.4 mg sublingual tablet) on Day 1.
- Zubsolv - Suboxone: Participants received Zubsolv® (buprenorphine 5.7 mg /naloxone 1.4 mg sublingual tablet) on Day 0 and Suboxone® (buprenorphine 8 mg /naloxone 2 mg sublingual film) on Day 1.
Period: Day 0 - First Treatment
Arm/Group | Suboxone - Zubsolv | Zubsolv - Suboxone
Started | 16 | 17
Completed | 15 | 16
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Day 1 - Second Treatment
Arm/Group | Suboxone - Zubsolv | Zubsolv - Suboxone
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- All Participants: Participants received Suboxone® (buprenorphine 8 mg /naloxone 2 mg sublingual film) on Day 0 and Zubsolv® (buprenorphine 5.7 mg /naloxone 1.4 mg sublingual tablet) on Day 1 or the reverse depending on randomized assignment.
Arm/Group | All Participants
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Intervention Preference As Assessed by Participants
Description: At the conclusion of Study Day 1, participants completed a study exit product comparison questionnaire. This outcome summarizes the percentage of participant answers to the question: When thinking about the two medications you evaluated over the last two days, which medication type did you prefer?
Time Frame: Day 1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
percentage of participants
  Suboxone | 54.84
  Zubsolv | 45.16
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p > 0.5000, Chi-squared — Two-tailed level of significance of 0.05 and no adjustments made for the number of tests conducted

2. Secondary Outcome: Participant Preference With Regard to Overall Taste of Interventions
Description: At the conclusion of Study Day 1, participants completed a study exit product comparison questionnaire. This outcome summarizes the percentage of participant answers to the question: Which one did you prefer in regards to overall taste?
Time Frame: Day 1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
percentage of participants
  Suboxone | 29.03
  Zubsolv | 70.97
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.0196, Chi-squared — Two-tailed level of significance of 0.05 and no adjustments made for the number of tests conducted

3. Secondary Outcome: Participant Assessments With Regard to Ease of Dissolution of Interventions
Description: At the conclusion of Study Day 1, participants completed a study exit product comparison questionnaire. This outcome summarizes the percentage of participant answers to the question: Which one did you think dissolve easier in your mouth?
Time Frame: Day 1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
percentage of participants
  Suboxone | 19.35
  Zubsolv | 80.65
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.0006, Chi-squared — Two-tailed level of significance of 0.05 and no adjustments made for the number of tests conducted

4. Secondary Outcome: Percentage of Participant Favorable and Unfavorable Response to the Question: How Easy or Difficult Was it to Open the Package?
Description: Responses were captured on a 5-point scale with the 5 representing the most favorable response, 3 representing a neutral response and 1 representing a negative response. 'Favorable' responses include assessments 5 and 4, while 'Unfavorable' responses include assessments 3, 2 and 1.
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 31 | 31
percentage of participants
  Favorable response | 61.29 | 51.61
  Unfavorable response | 38.71 | 48.39
Statistical Analysis 1: Comparison: Suboxone Sublingual Film 8/2 vs Zubsolv Sublingual Tablets 5.7/1.4; Test type: Superiority or Other; p = 0.4422, Chi-squared — Two-tailed level of significance of 0.05 and no adjustments made for the number of tests conducted

5. Secondary Outcome: Percentage of Participant Favorable and Unfavorable Response to the Question: How Easy or Difficult Were the Package Instructions to Follow?
Description: as for outcome 4
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 30 | 31
percentage of participants
  Favorable response | 100 | 90.32
  Unfavorable response | 0 | 9.68
Statistical Analysis 1: Comparison: Suboxone Sublingual Film 8/2 vs Zubsolv Sublingual Tablets 5.7/1.4; Test type: Superiority or Other; p = 0.2377, Chi-squared

6. Secondary Outcome: Percentage of Participant Favorable and Unfavorable Response to the Question: How Comfortable Did It Feel In Your Mouth?
Description: as for outcome 4
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 31 | 31
percentage of participants
  Favorable response | 54.84 | 77.42
  Unfavorable response | 45.16 | 22.58
Statistical Analysis 1: Comparison: Suboxone Sublingual Film 8/2 vs Zubsolv Sublingual Tablets 5.7/1.4; Test type: Superiority or Other; p = 0.0603, Chi-squared

7. Secondary Outcome: Percentage of Participant Favorable and Unfavorable Response to the Question: How Easily Did the Medication Dissolve in Your Mouth?
Description: as for outcome 4
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 31 | 31
percentage of participants
  Favorable response | 54.84 | 96.77
  Unfavorable response | 45.16 | 3.23
Statistical Analysis 1: Comparison: Suboxone Sublingual Film 8/2 vs Zubsolv Sublingual Tablets 5.7/1.4; Test type: Superiority or Other; p < 0.0010, Chi-squared

8. Secondary Outcome: Percentage of Participant Response to the Question: Did You Experience Any Uncomfortable Effects of Burning or Stinging?
Description: Participant responses were captured on a 10-point scale with 0 = None and 9= Extreme.
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 31 | 31
percentage of participants
  0 (none) | 67.74 | 58.06
  1 | 19.35 | 19.35
  2 | 6.45 | 16.13
  3 | 3.23 | 0
  4 | 0 | 0
  5 | 3.23 | 3.23
  6 | 0 | 0
  7 | 0 | 0
  8 | 0 | 0
  9 (extreme) | 0 | 3.23

9. Secondary Outcome: Percentage of Participant Response to the Question: Did You Experience Any Uncomfortable Effects of Skin Irritation or Blisters?
Description: Participant responses were captured on a 10-point scale with 0 = None and 9= Extreme.
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 31 | 31
percentage of participants
  0 (none) | 70.97 | 70.97
  1 | 22.58 | 29.03
  2 | 3.23 | 0
  3 | 0 | 0
  4 | 0 | 0
  5 | 3.23 | 0
  6 | 0 | 0
  7 | 0 | 0
  8 | 0 | 0
  9 (extreme) | 0 | 0

10. Secondary Outcome: Percentage of Participant Response to the Request: Please Rate the Medication You Received Today in Terms of the Drug's Ability to Product a 'High'
Description: Participant responses were captured on a 10-point scale with 0 = No high and 9= Extremely strong high.
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 31 | 31
percentage of participants
  0 (no high) | 70.97 | 61.29
  1 | 16.13 | 32.26
  2 | 9.68 | 6.45
  3 | 0 | 0
  4 | 0 | 0
  5 | 3.23 | 0
  6 | 0 | 0
  7 | 0 | 0
  8 | 0 | 0
  9 (extremely strong high) | 0 | 0

11. Secondary Outcome: Percentage of Participant Response to the Request: When Thinking About the Medication You Used Today, Indicate on the Line Below Your Ability to Abuse This Medication
Description: Participant responses were captured on a 10-point scale with 0 = No desire to abuse and 9= Extremely high desire to abuse.
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 31 | 31
percentage of participants
  0 (no high) | 70.97 | 61.29
  1 | 16.13 | 35.48
  2 | 9.68 | 3.23
  3 | 0 | 0
  4 | 0 | 0
  5 | 3.23 | 0
  6 | 0 | 0
  7 | 0 | 0
  8 | 0 | 0
  9 (extremely strong high) | 0 | 0

12. Secondary Outcome: Percentage of Participant Response to the Question: If You Did Want to Abuse This Medication, Would You Prefer to......
Description: Choices to the question above are:
  * Crush and snort
  * Liquefy and inject
  * Not able to abuse this formulation
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 31 | 31
percentage of participants
  Crush and snort | 0 | 25.81
  Liquefy and inject | 0 | 3.23
  Not able to abuse this formulation | 100 | 70.97

13. Secondary Outcome: Percentage of Participant Response to the Question: Compared to the Medication That You Are Currently Using for Treatment of Opioid Dependence, The Study Medication You Just Used Was.....
Description: Choices to the question above are:
  * More effective as a treatment for opioid dependence
  * Equally effective as a treatment for opioid dependence
  * Less effective as a treatment for opioid dependence
  * The same medication that I normally use
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 31 | 31
percentage of participants
  More effective | 3.23 | 0
  Equally effective | 29.03 | 51.61
  Less effective | 0 | 32.26
  Same medication I normally use | 67.74 | 16.13

14. Secondary Outcome: Dissolution Time of Intervention as Recorded by a Trained Observer
Description: The subject was observed and times documented for time of administration and time dissolution (recorded in minutes and seconds) was completed by designated qualified study personnel at the site.
Time Frame: Days 0-1
Population: The per-protocol population included participants who did not miss any visit and had no major protocol violations.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 32 | 32
minutes | 6.59 (5.28) | 2.98 (2.48)

15. Secondary Outcome: Change From Baseline in Subject Opiate Withdrawal Scale (SOWS)
Description: Participants completed the Subject Opiate Withdrawal Scale (SOWS) at baseline, and the end of each day of treatment.
  SOWS is a validated scale when used as defined. The research site did not use SOWS as defined. The sponsor made the decision to not report this data since it was not captured in a validated format.
Time Frame: Day 0 prior to dosing, end of Day 0 (post dose), end of Day 1 (post dose)
Population: Per protocol set.
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Days 0 (post treatment) -1
Arm/Group | Suboxone Sublingual Film 8/2 | Zubsolv Sublingual Tablets 5.7/1.4
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 3/32 | 13/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suboxone Sublingual Film 8/2 (N=32) | Zubsolv Sublingual Tablets 5.7/1.4 (N=32)
Rhinnorhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 2 | 8
Constipation (Gastrointestinal disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multi-center publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.